CLINICAL TRIAL: NCT00065572
Title: Exploratory Study to Assess the Biological Activity of ZD6126 in Subjects With Newly Diagnosed Metastatic Renal Cell Carcinoma (Stage IV)
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D2820C00018; 6126IL/00018
Record Dates: First submitted 2003-07-28; First posted 2003-07-31 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Carcinoma, Renal Cell; Kidney Neoplasms
Keywords: Kidney Cancer; Metastatic; Newly diagnosed renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Neoplasm Metastasis | interventions — N-acetylcochinol-O-phosphate

INTERVENTIONS:
Drug: ZD6126
Drug: Placebo

SUMMARY:
The purpose of this study is to assess the biological activity of ZD6126 in subjects with newly diagnosed metastatic renal cell carcinoma (stage IV).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed metastatic renal cell carcinoma
* Suitable for nephrectomy

Exclusion Criteria:

* Prior chemotherapy, biological therapy or radiation therapy for renal cell carcinoma or within the last 3 years for any other cancer
* Significant cardiac event within 3 months of entry
* Any history of coronary angioplasty or history of myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-08; Primary Completion 2004-02 (Estimated); Study Completion 2004-02 (Estimated)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Research Site, Los Angeles, California
  - Research Site, Newark, Delaware
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Baltimore, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, Lebanon, New Hampshire
  - Research Site, Hackensack, New Jersey
  - Research Site, Rochester, New York
  - Research Site, The Bronx, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Salt Lake City, Utah